CLINICAL TRIAL: NCT05765799
Title: Evaluation of Patient Information in Interventional Radiology.
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1482021/CHUSTE
Record Dates: First submitted 2023-02-27; First posted 2023-03-13 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Patient Satisfaction
Keywords: interventional radiology; Information; videos
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient who receives a consultation before an interventional procedure: Any patient who receives a consultation before an interventional procedure will be included. Questionary will be administrated.
  Interventions: Other: Questionary

INTERVENTIONS:
Other: Questionary — Questionary will be administrated to evaluated the information for patients on interventional radiology (dedicated consultation, information posters, explanatory video, information form, etc.).

SUMMARY:
Interventional radiology is developing. Patient information modalities are also evolving, in particular information videos.

The aim of this work is therefore the evaluation of patient information in interventional radiology

ELIGIBILITY:
Inclusion Criteria:

* Any patient who receives a consultation before an interventional procedure.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who receives a consultation before an interventional procedure will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate effectiveness of each patient information tool by Consultation with the interventional radiologist | Year : 2
  Analysis results of questionary.
To evaluate Effectiveness of each patient information tool by Consultation with another doctor who explained the procedure | Year : 2
  Analysis results of questionary.
To evaluate Effectiveness of each patient information tool by Explanatory videos | Year : 2
  Analysis results of questionary.
To evaluate Effectiveness of each patient information tool by Patient information sheet | Year : 2
  Analysis results of questionary.
To evaluate Effectiveness of each patient information tool by Posters in the consultation room | Year : 2
  Analysis results of questionary.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain GRANGE, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No